CLINICAL TRIAL: NCT05088187
Title: Longitudinal Evaluation of Objective Cognitive Function and Quality of Life in Patients Undergoing Surgery for Malignant and Benign Thyroid Nodules
Brief Title: Cognition and QoL After Thyroid Surgery
Status: Recruiting | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: The Netherlands Cancer Institute (Other)
Responsible Party: Principal Investigator, Renske Altena, MD PhD, Karolinska University Hospital
Other Study IDs: CogniThyr
Record Dates: First submitted 2021-10-11; First posted 2021-10-21 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Thyroid Nodule; Thyroid Cancer; Cognitive Decline; Survivorship; Symptoms, Cognitive
MeSH Terms: conditions — Thyroid Nodule; Thyroid Neoplasms; Cognitive Dysfunction; Neurobehavioral Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The development of cognitive dysfunction can profoundly affect HR-QoL as well as the possibility of societal participation and ability to work, and thereby relevantly impacts prospects for cancer survivorship. The aim of the study is to obtain improved understanding of the scope and magnitude of objective cognitive dysfunction in DTC survivors, and its relation to subjective cognitive dysfunction, thyroid hormone levels, physical activity and HRQoL. This is done in a prospective study where patients operated for a thyroid nodule (Bethesda IV-VI, i.e., benign [goitre with nodule and fibroadenomas], low-risk DTC and intermediate-high risk DTC) are included and asked to serially perform online neuropsychological testing as well as to complete questionnaires related to HR-QoL, physical activity and additional psychological and physical complaints. Blood is analysed for levels of thyroid hormones and systemic inflammation.

DETAILED DESCRIPTION:
The primary aim of this study is to prospectively assess objective cognitive functioning in patients undergoing thyroid surgery for different indications by means of an online neuropsychological test, the Amsterdam Cognition Scale (ACS).

Three patient groups are defined; 1) patients with follicular adenomas, 2) patients with extreme low-risk differentiated thyroid cancer (DTC; pT1a and pN0/x tumours), 3) patients in all other DTC risk groups (i.e., low, intermediate and high-risk). The primary comparison confers to groups 1 and 3.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old, indication for surgery because of a thyroid nodule Bethesda IV-VI
* Able to read and understand the Swedish language
* Access to desktop computer or laptop with internet connection
* Able and willing to provide written informed consent

Exclusion Criteria:

* A previous diagnosis of (auto-immune) hypothyroidism
* A previous cancer diagnosis (excluding basal cell cancer of the skin)
* Indications for surgery other than (solely) a thyroid nodule (i.e., concomitant Graves)
* A diagnosis of medullary and anaplastic thyroid cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who are visiting the Medical Unit Endocrine Tumours at the Karolinska University Hospital and scheduled for thyroid surgery for Bethesda IV-VI thyroid lesions, will be informed about the possibility to participate in this study.
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Objective cognitive functioning by means of an online neuropsychological test (Amsterdam Cognition Scale, ACS) | pre-surgery to 12 months post-surgery
  change in total score on ACS

CONTACTS AND LOCATIONS:
Overall Officials: Renske Altena, MD PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Medical Unit Breast-, Endocrine tumors and Sarcoma, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share IPD upon request directly to the investigators